CLINICAL TRIAL: NCT03132922
Title: Phase 1 Dose Escalation, Multi-tumor Study to Assess the Safety, Tolerability and Antitumor Activity of Genetically Engineered MAGE-A4ᶜ¹º³²T in HLA-A2+ Subjects With MAGE-A4 Positive Tumors
Brief Title: MAGE-A4ᶜ¹º³²T for Multi-Tumor
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0044-001/RSS
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Urinary Bladder Cancer; Melanoma; Head and Neck Cancer; Ovarian Cancer; Non-Small Cell Lung Cancer; Esophageal Cancer; Gastric Cancer; Synovial Sarcoma; Myxoid Round Cell Liposarcoma; Gastroesophageal Junction
Keywords: Cell Therapy; T Cell Therapy; SPEAR T Cell; MAGE-A4; Immuno-oncology; Metastatic; Urothelial Cancer; Previously Treated; T Cell Receptor; Squamous, adenosquamous, adenocarcinoma or large cell NSCLC; Squamous or adenocarcinoma esophageal cancer; Sarcoma; Melanoma; Bladder; Ovarian; Radiation therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Melanoma; Head and Neck Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Stomach Neoplasms; Sarcoma, Synovial; Liposarcoma, Myxoid; Neoplasm Metastasis; Adenocarcinoma; Sarcoma | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Autologous genetically modified MAGE-A4ᶜ¹º³²T cells (Experimental)
  Interventions: Genetic: Autologous genetically modified MAGE-A4ᶜ¹º³²T cells
- Radiation Sub-Study: Autologous genetically modified MAGE-A4c1 (Experimental)
  Interventions: Radiation: Autologous genetically modified MAGE-A4c1032T cells combined with low dose radiation

INTERVENTIONS:
Genetic: Autologous genetically modified MAGE-A4ᶜ¹º³²T cells — Infusion of autologous genetically modified MAGE-A4ᶜ¹º³²T on Day 1
  Arms: Autologous genetically modified MAGE-A4ᶜ¹º³²T cells
Radiation: Autologous genetically modified MAGE-A4c1032T cells combined with low dose radiation — Up to 10 subjects will be considered for Radiation sub-study. Radiation with an intensity of 1.4Gy for 5 days before infusion of MAGE-A4c1032T cells
  Arms: Radiation Sub-Study: Autologous genetically modified MAGE-A4c1

SUMMARY:
This study will investigate the safety and tolerability of MAGE-A4ᶜ¹º³²T cell therapy in subjects who have the appropriate HLA-A2 tissue marker and whose urinary bladder, melanoma, head and neck, ovarian, non-small cell lung, esophageal, gastric, synovial sarcoma, or myxoid/round call liposarcoma (MRCLS) tumor has the MAGE-A4 protein expressed. This study will take a subject's T cells and give them a T cell receptor protein that recognizes and attacks the tumors. This study has a substudy component that will investigate the safety and tolerability of MAGE-A4c1032T cell therapy in combination with low dose radiation in up to 10 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 to 75 years of age at the time of signing the study informed consent.
2. Subject has histologically confirmed diagnosis of any one of the indicated tumor types
3. Subject is HLA-A*02 positive. (This determination will be made under screening protocol ADP-0000-001).
4. Subject's tumor shows expression of the MAGE-A4 RNA or protein. (This determination will be made under screening protocol ADP-0000-001).
5. Adequate organ function as indicated in the study protocol
6. Subject has measurable disease according to RECIST v1.1 criteria prior to lymphodepletion
7. Subject meets disease-specific requirements per protocol

7. Subject has anticipated life expectancy > 6 months prior to leukapheresis and >3 months prior to lymphodepletion.

Exclusion Criteria:

1. Subject does not express appropriate HLA-A genotype
2. Subject is receiving excluded therapy/treatment per protocol
3. Subject has symptomatic CNS metastases.
4. Subject has any other active malignancy besides the tumor under study within 3 years prior to Screening. Subject has uncontrolled intercurrent illness.
5. Subject has active infection with HIV, HBV, HCV or HTLV
6. Subject is pregnant or breastfeeding.

Additional Exclusion Criteria for the Radiation Substudy:

* Subject does not meet eligibility criteria for the main study (ADP-0044-001).
* Subject does not have at least one target lesion amenable to radiation.
* Certain radiation therapy within 6 months of clinical trial are an exclusion.
* Metastatic disease impinging on the spinal cord or threatening spinal cord compression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AE), including serious adverse events (SAEs). | 3.5 years
  Determine if treatment with autologous genetically modified T cells (MAGE-A4ᶜ¹º³²T) is safe and tolerable through laboratory assessments including chemistry, hematology and coagulation.
Determining dose limiting toxicities (DLT) and optimally tolerated dose range | 3.5 years
  Evaluate DLTs and toxicity assessment using NCI CTCAE.
Evaluation of persistence of genetically modified T cells. | 3.5 years
  Evaluation of persistence of genetically modified T cells in the periphery.
Measurement of RCL in genetically modified T cells. | 3.5 years
  Evaluation of RCL in subject PBMCs using PCR-based assay.

SECONDARY OUTCOMES:
Proportion of subjects with a confirmed Complete Response (CR) and/or Partial Response (PR). | 3.5 years
  Evaluation of the efficacy of the treatment by assessment of the Overall Response Rate according to RECIST v1.1
Interval between the date of first T cell infusion dose and first documented evidence of CR or PR. | 3.5 years
  Evaluation of the efficacy of the treatment by assessment of time to first response.
Interval between the date of first documented evidence of CR or PR until first documented disease progression or death due to any cause. | 3.5 years
  Evaluation of the efficacy of the treatment by assessment of duration of response.
Interval between the date of first documented evidence of stable disease (SD) until first documented disease progression or death due to any cause. | 3.5 years
  Evaluation of the efficacy of the treatment by assessment of duration of stable disease.
Interval between the date of first T cell infusion and the earliest date of disease, progression or death due to any cause | 3.5 years
  Evaluation of the efficacy of the treatment by assessment of progression-free survival.
Interval between the date of first T cell infusion and date of death due to any cause. | 3.5 years
  Evaluation of the efficacy of the treatment by assessment of overall survival.
Number and % of subjects having any Long Term Follow Up Adverse Events (AEs) | 15 years post last treatment (infusion)
  * New occurrence of any malignancy
  * New occurrence or exacerbation of a pre-existing neurologic disorder
  * New occurrence or exacerbation of a prior rheumatologic or other autoimmune disorder
  * New occurrence of a hematologic disorder
  * New occurrence of any opportunistic and/or serious infections
  * New occurrence of any unanticipated illness and/or hospitalization deemed related to gene modified cell therapy

OTHER OUTCOMES:
MAGE-A4c1032T cell trafficking in tumor lesion(s). | 3.5 years
  Evaluation of post-infusion T-cell trafficking in irradiated vs non-irradiation lesions

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (11):
- United States (10):
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Duke Cancer Institute, Durham, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology - Sarah Cannon Research Institute, Nashville, Tennessee
  - M.D. Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Hong DS, Van Tine BA, Biswas S, McAlpine C, Johnson ML, Olszanski AJ, Clarke JM, Araujo D, Blumenschein GR Jr, Kebriaei P, Lin Q, Tipping AJ, Sanderson JP, Wang R, Trivedi T, Annareddy T, Bai J, Rafail S, Sun A, Fernandes L, Navenot JM, Bushman FD, Everett JK, Karadeniz D, Broad R, Isabelle M, Naidoo R, Bath N, Betts G, Wolchinsky Z, Batrakou DG, Van Winkle E, Elefant E, Ghobadi A, Cashen A, Grand'Maison A, McCarthy P, Fracasso PM, Norry E, Williams D, Druta M, Liebner DA, Odunsi K, Butler MO. Autologous T cell therapy for MAGE-A4+ solid cancers in HLA-A*02+ patients: a phase 1 trial. Nat Med. 2023 Jan;29(1):104-114. doi: 10.1038/s41591-022-02128-z. Epub 2023 Jan 9. PMID 36624315
- [Derived] Sanderson JP, Crowley DJ, Wiedermann GE, Quinn LL, Crossland KL, Tunbridge HM, Cornforth TV, Barnes CS, Ahmed T, Howe K, Saini M, Abbott RJ, Anderson VE, Tavano B, Maroto M, Gerry AB. Preclinical evaluation of an affinity-enhanced MAGE-A4-specific T-cell receptor for adoptive T-cell therapy. Oncoimmunology. 2019 Nov 24;9(1):1682381. doi: 10.1080/2162402X.2019.1682381. eCollection 2020. PMID 32002290